CLINICAL TRIAL: NCT06484829
Title: An Open-Label, Parallel-Controlled, Multi-Center Phase Ib/IIa Clinical Study to Evaluate the Efficacy and Safety of Purinostat Mesylate for Injection Combined With Pomalidomide Capsules and Low-Dose Dexamethasone in Patients With Relapsed and Refractory Multiple Myeloma
Brief Title: Purinostat Mesylate Combined With Pomalidomide Capsules and Low-dose Dexamethasone in Patients With Relapsed or Refractory Multiple Myeloma
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Chengdu Zenitar Biomedical Technology Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: ZLPM-002-1.0
Record Dates: First submitted 2024-05-21; First posted 2024-07-03 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-03

CONDITIONS: Relapsed or Refractory Multiple Myeloma (RRMM)
MeSH Terms: conditions — Recurrence; Multiple Myeloma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- A group (Experimental): A: Treatment Cycle Regimen - Regimen A (2-Week On/1-Week Off) - 21-Day Cycle
  Purinostat Mesylate for Injection: Intravenous infusion on Days 1, 4, 8, and 11 of each 21-day (3-week) cycle during the Continuation Dosing Phase Ib and Phase IIa;
  Pomalidomide Capsules: Oral administration once daily at 4 mg for 14 consecutive days followed by a 7-day rest period, with each cycle lasting 21 days (3 weeks);
  Dexamethasone Acetate Tablets: 20 mg orally administered on Days 1, 4, 8, and 11 of each treatment cycle.
  Interventions: Drug: Purinostat Mesylate 4 mg/m2; Drug: Purinostat Mesylate 6 mg/m2; Drug: Purinostat Mesylate 8.4 mg/m2
- B group (Experimental): B: Treatment Cycle Regimen - Regimen B (3-Week On/1-Week Off) - 28-Day Cycle
  Purinostat Mesylate for Injection: Intravenous infusion on Days 1, 4, 15, and 18 of each 28-day (4-week) cycle during the Continuation Dosing Phase 1b and Phase IIa;
  Pomalidomide Capsules: Oral administration once daily at 4 mg for 21 consecutive days followed by a 7-day rest period, with each cycle lasting 28 days (4 weeks);
  Dexamethasone Acetate Tablets: 20 mg orally administered on Days 1, 4, 15,and 18 of each treatment cycle.
  Interventions: Drug: Purinostat Mesylate 4 mg/m2; Drug: Purinostat Mesylate 6 mg/m2; Drug: Purinostat Mesylate 8.4 mg/m2

INTERVENTIONS:
Drug: Purinostat Mesylate 4 mg/m2 — 4 mg/m2 Purinostat Mesylate + 4mg Pomalidomide + 20mg Dexamethasone.
Drug: Purinostat Mesylate 6 mg/m2 — 6 mg/m2 Purinostat Mesylate + 4mg Pomalidomide + 20mg Dexamethasone.
Drug: Purinostat Mesylate 8.4 mg/m2 — 8.4 mg/m2 Purinostat Mesylate + 4mg Pomalidomide + 20mg Dexamethasone.

SUMMARY:
Primary Purpose Phase Ib. To determine the Maximum Tolerated Dose (MTD) and establish the Recommended Phase IIa Dose (RP2D) of Purinostat Mesylate for Injection combined with fixed-dose Pomalidomide Capsules and Dexamethasone in patients with relapsed or refractory multiple myeloma.

Phase IIa. To further evaluate the safety and tolerability of Purinostat Mesylate for Injection at the RP2D combined with fixed-dose Pomalidomide Capsules and Dexamethasone in patients with relapsed and refractory multiple myeloma (RRMM).

Secondary Objectives Phase Ib

1. To evaluate the safety and tolerability of Purinostat Mesylate for Injection combined with fixed-dose Pomalidomide Capsules and Dexamethasone in the treatment of relapsed or refractory multiple myeloma.
2. To assess the pharmacokinetic (PK) parameters of the combination therapy in patients with relapsed or refractory multiple myeloma.
3. To observe the preliminary efficacy of the combination therapy in patients with relapsed or refractory multiple myeloma.

Phase IIa

1. To evaluate the preliminary efficacy of the combination therapy in patients with relapsed and refractory multiple myeloma (RRMM).
2. To characterize the population pharmacokinetic (PPK) profile of the combination therapy in patients with relapsed or refractory multiple myeloma (RRMM).

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed with multiple myeloma (MM) by reference to the diagnostic criteria of the Chinese Guidelines for the Diagnosis and Treatment of Multiple Myeloma (Revised 2022);
2. Those who have received at least one line of prior systemic antimyeloma therapy (which must include lenalidomide and proteasome inhibitors; see Appendix 4 for counts of myeloma treatment lines) and meet the definition of relapse or refractory; Definition of relapse: disease progression that occurs at least 60 days from the last treatment after the efficacy of a prior treatment regimen was evaluated at MR or better (except for those who relapsed more than 1 year after treatment); Definition of refractory: progression during prior therapy or progression within 60 days of the last treatment; or failure to achieve MR or better after at least 2 prior courses of therapy; or treatment intolerance.
3. Age 18-75 years, male or female, if of childbearing potential subjects should be on effective contraception and must agree to comply with all contraceptive requirements:

1) Females of childbearing potential must agree to and comply with the contraceptive measures specified in the protocol: beginning 4 weeks prior to treatment with this product, two reliable methods of contraception are required concurrently for the duration of the treatment, during the dose suspension, and for 4 weeks after termination of the treatment (one highly effective method of contraception-tubal ligation, intrauterine device, hormonal (contraceptive pills, injections, patches, vaginal rings, or implants), or partner's vasectomy, and another effective contraceptive method - male rubber or synthetic condom, diaphragm or cervical cap). Effective contraception is needed even with a history of infertility unless due to hysterectomy; 2) Men of childbearing potential must use a rubber or synthetic condom at all times during sexual contact with women of childbearing potential beginning 4 weeks prior to treatment with this product, during the treatment period, during the dose suspension period, and for 4 weeks after termination of treatment, even if they have had a successful vasectomy; 4. Subjects with multiple myeloma who have measurable M protein, i.e., at least one of the following 3 measurements:

1. Serum M protein ≥ 0.5 g/dL (5 g/L);
2. Urine M protein ≥ 200 mg/24h;
3. Serum free light chain assay: in the case of an abnormal serum free light chain ratio (less than 0.26 or greater than 1.65), an affected free light chain level ≥10mg/dL (100mg/L); 5. Hematologic fulfillment of the following conditions:

1) ANC ≥ 1.0 x 109/L (without granulocyte colony-stimulating factor within 7 days), with no specific requirement for neutrophil count when ≥ 50% of the bone marrow is plasma cells; 2) PLT ≥75 × 109/L (no platelet transfusion or use of thrombopoietin within 7 days), and platelets ≥50 × 109/L were eligible for enrollment when ≥50% of plasma cells were present in the bone marrow; 3) Hemoglobin ≥ 80 g/L (no red blood cell suspension infusion or use of erythropoietin within 7 days); 6. Liver and kidney function tests fulfill the following conditions:

1. TBIL ≤ 1.5 x ULN;
2. ALT and AST are ≤ 2.5 x ULN;
3. Glomerular filtration rate (GFR) ≥ 30mL/min/1.73m2 (Cockcroft-Gault formula) without the effects of dialysis therapy; 7. Ability to receive and have access to antithrombotic medications such as low molecular heparin sodium, heparin, warfarin or aspirin; 8. An ECOG (Appendix 2) score of 0-2 and an expected survival of ≥12 weeks; 9. Subjects voluntarily enrolled in the study and signed an informed consent form.

Exclusion Criteria:

1. Those with prior antitumor therapy with histone deacetylase (HDAC) inhibitors (except cedarbenazine), antibody-coupled degradation agents (DAC), HSP90 inhibitors, or valproic acid; or those who, in the judgment of the investigator, are intolerant to treatment with the same type of drug as HDAC inhibitors, pomalidomide, thalidomide, lenalidomide, or the like (e.g., grade ≥3 rash during prior use, severe refractory myelosuppression, etc.);
2. Those with disease progression following prior treatment with standard dose pomalidomide;
3. Allergic reactions to the components of the test drug involved in this trial;
4. A diagnosis of non-secretory MM (defined as a subject who is completely non-secretory or who has a small amount of free light chain but the affected light chain is less than 100 mg/L), or MM in combination with amyloidosis, or plasma cell leukemia, either primary or during the course of therapy
5. Those with active new thrombosis or who are unable to receive antithrombotic therapy;
6. Other malignant tumors within 5 years prior to screening, with the exception of cured carcinoma in situ (e.g., cervix, breast, bladder, etc.), basal cell carcinoma of the skin, squamous epithelial cell carcinoma of the skin, or early-stage prostate carcinoma (with clinical staging of Tla or T1b);
7. Those who have a combination of central nervous system disorders and require treatment for such disorders
8. Peripheral neuropathy ≥ grade 3; and
9. Co-morbidities requiring long-term treatment with immunosuppressive drugs or steroids; 10. active infectious diseases;
10. Those with comorbid active infectious diseases, including the following:

1) Hepatitis B Surface Antigen (HbsAg) or Hepatitis B Core Antibody (HbcAb) positive with HBV-DNA quantification higher than the upper limit of normal value 2) Positive Hepatitis C Virus Antibody (HCV-Ab) with HCV RNA quantification above the upper limit of normal; 3) Human immunodeficiency virus antibody (HIV-Ab) or anti-syphilis spirochete antibody (TP-Ab) positive; 11. Subjects with any of the following:

1. Cardiac insufficiency ≥ grade 3 by NYHA classification (Appendix 1) criteria;
2. Myocardial infarction within 6 months;
3. Poorly controlled angina, including variant angina, within 6 months;
4. Clinically significant arrhythmia;
5. ECG QTcF >450 ms (men) and QTcF >470 ms (women) (Fridericia formula);
6. Echocardiographic indication of left ventricular ejection fraction <50%; 12. A combination of severe infectious disease requiring systemic intravenous antibiotic therapy 2 weeks prior to the first dose; 13. Those who have received an allogeneic hematopoietic stem cell transplant within 12 months, or those who have active graft-versus-host disease (GVHD) or GVHD requiring immunosuppressive therapy more than 12 months after the allogeneic hematopoietic stem cell transplant; 14. Who have participated in another clinical trial within 4 weeks prior to the first dose; 15. Those who have received other antitumor therapy (including herbal antitumor therapy, except for ≤20 mg/day of prednisone and its equivalent dose of steroid hormones) within 2 weeks prior to the first administration of the drug; 16. Those who have not recovered to Grade 1 or below from toxic reactions to prior antitumor therapy (except alopecia, malaise and those limited by entry criteria #6); 17. Those who have received major surgical treatment within 4 weeks prior to the first dose and have not fully recovered; 18. Women who are pregnant or breastfeeding; 19. Persons who, in the opinion of the investigator, have other factors that make them unsuitable for participation in the trial (e.g., uncontrolled active hypertension, uncontrolled active diabetes mellitus, poor adherence, substance abuse, etc.).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Estimated)
Dates: Start 2024-03-25 (Actual); Primary Completion 2026-02-01 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
Dose-limiting toxicity (DLT) | Day 21/Day 28
  One or more unacceptable toxic reactions following administration of the drug, resulting in the inability to continue increasing the dose or prolonging the dosing cycle
Maximum Tolerated Dose (MTD) | Day 21/Day 28
  The maximum dose or concentration of a drug that does not cause death in experimental animals in experiments other than acute toxicity animal experiments (short-term repetitive experiments, subchronic toxicity experiments, chronic toxicity experiments).
Objective remission rate (ORR) | Day 21/Day 28
  Defined as the proportion of subjects achieving a strict complete remission (sCR) + complete remission (CR) + very good partial remission (VGPR) + partial remission (PR);

SECONDARY OUTCOMES:
Complete Remission Rate (CRR) | Day 21/Day 28
  Proportion of subjects with sCR+CR
Duration of efficacy (DOR) | Day 21/Day 28
  Duration of first remission (PR and above) to disease progression or death;
Time to Relief (TTR) | Day 21/Day 28
  Time from first dose to PR and beyond
Progression-free survival (PFS) | Day 21/Day 28
  Time from first dose to disease progression or death
Overall survival (OS) | Day 21/Day 28
  Time from first dose to death from all causes

CONTACTS AND LOCATIONS:
Overall Officials: Ting Niu, Doctor, Principal Investigator — West China Hospital
Locations (1):
- West China Hospital Sichuan University, Chengdu, Sichuan, China